CLINICAL TRIAL: NCT05246228
Title: Immune System Modulation and Outcome in High-risk Cutaneous Squamous Cell Carcinoma Treated With Surgery and Radiotherapy: a Prospective Study
Brief Title: Immune System Modulation and Outcome in High-risk cSCC Treated With Surgery and Radiotherapy
Acronym: HR-cSCC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Collaborators: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); Azienda Ospedaliera di Padova (Other); Istituti Ospitalieri di Cremona (Other); IRCCS Sacro Cuore Don Calabria di Negrar (Other); ASST Bergamo Ovest (Other); San Gerardo Hospital (Other); ASST Valcamonica (Unknown)
Responsible Party: Principal Investigator, Paolo Bossi, Clinical Professor, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Other Study IDs: ASST Spedali Civili di Brescia
Record Dates: First submitted 2021-11-25; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Squamous Cell Carcinoma of the Skin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with cSCC addressed to adjuvant radiotherapy as per clinical practice: The aim of the study is to evaluate patient's outcome according to the post-radiation lymphocytes count and to the changes induced in the immune cell population by a loco-regional treatment as radiotherapy. The way to objectivate these results is to collect some blood samples and analyze them.
  Interventions: Other: Peripheral blood sampling in order to evaluate changes in the circulating immune population

INTERVENTIONS:
Other: Peripheral blood sampling in order to evaluate changes in the circulating immune population — Eveluation: circulating T cells CD3+CD8+ and CD3+CD4+, absolute lymphocyte count (ALC) and neutrophil counts (ANC) and neutrophil/lymphocyte ratio (NLR), Treg lymphocytes, Naïve/Memory T lymphocytes CD4+ and CD8+,myeloid-derived suppressor cells, Plasmacytoid Dendritic Cells NK cells dimension and bright, NKT cells, Myeloid Dendritic cells, Monocytes subsets, B lymphocytes ,Analysis of plasma cytokines (TNFalpha, TGFbeta, IL-6, IL-10) by ELISA,FN signature: real-time PCR on mRNA from peripheral blood mononuclear cells (PBMCs)

SUMMARY:
Treatment with adjuvant radiotherapy modulates immune system in many diseases as witnessed by dynamic changes of humoral and cellular immunity. Moreover, the persistent lymphopenia after radiation therapy is a negative prognostic factor. This study is aimed to explore the changes in immune-cell populations during radiotherapy given as adjuvant treatment for high-risk cutaneous squamous cell carcinomas and to correlate them with patient's outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Signed written informed consent.
* Histologically confirmed diagnosis of cSCC.
* cSCC categorized as high risk according to ASTRO Guidelines:

  * close or positive margins that cannot be corrected with further surgery (secondary to morbidity or adverse cosmetic outcome).
  * gross perineural spread, as identified by radiological or pathological assessment.
  * disease recurrence after a prior margin-negative resection.
  * pathological stage T3 and T4.
  * desmoplastic or infiltrative tumors in the setting of chronic immunosuppression at pathological exam, cSCC involving regional lymphnodes, with the exception of a single, small (<3 cm) cervical lymph node harboring carcinoma, without extracapsular extension.
* cSCC addressed to adjuvant radiotherapy as per clinical practice (a complete post-operative treatment should be administered with 50-54 or 60-66 Gy depending on the margin status).
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0-2.

Exclusion Criteria:

* cSCC not eligible for surgery.
* cSCC not eligible for adjuvant radiotherapy for any condition depending on disease characteristics or patient characteristics, co-morbidities or refusal.
* Any concurrent investigational product, biologic, or hormonal therapy for cancer treatment.
* Concurrent treatment with chemotherapy for the purpose of cSCC cure.
* History or current evidence of any condition that, in the opinion of the treating investigator, might interfere with the subject's participation for the full duration of the trial.
* Any major surgery, different from that planned for the protocol, in the 15 days before the protocol starting.
* Any radiotherapy treatment in the 28 days before the protocol starting
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients enrolled in the study are affected form cSCC classified at high risk and addressed to surgery and subsequent adjuvant radiotherapy according to clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) of patients with ALC < 500 cells/mL 28 days after the end of radiotherapy treatment | 28 days after the end of radiotherapy treatment
  Disease-free survival (DFS) of patients with ALC < 500 cells/mL 28 days after the end of radiotherapy treatment

SECONDARY OUTCOMES:
Evaluation of changes (Δ) in the circulating immune-cells population before the start of radiotherapy and 28 days after the end of radiotherapy | Before and 28 days after the end of radiotherapy treatment
  Evaluation of changes (Δ) in the circulating immune-cells population before the start of radiotherapy and 28 days after the end of radiotherapy.
  Correlation between DFS and circulating immune cell population

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bossi, MD, Principal Investigator — ASST Spedali Civili

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lin AJ, Gang M, Rao YJ, Campian J, Daly M, Gay H, Oppelt P, Jackson RS, Rich J, Paniello R, Zevallos J, Hallahan D, Adkins D, Thorstad W. Association of Posttreatment Lymphopenia and Elevated Neutrophil-to-Lymphocyte Ratio With Poor Clinical Outcomes in Patients With Human Papillomavirus-Negative Oropharyngeal Cancers. JAMA Otolaryngol Head Neck Surg. 2019 May 1;145(5):413-421. doi: 10.1001/jamaoto.2019.0034. PMID 30920592
- [Result] Que SKT, Zwald FO, Schmults CD. Cutaneous squamous cell carcinoma: Incidence, risk factors, diagnosis, and staging. J Am Acad Dermatol. 2018 Feb;78(2):237-247. doi: 10.1016/j.jaad.2017.08.059. PMID 29332704
- [Result] Stratigos AJ, Garbe C, Dessinioti C, Lebbe C, Bataille V, Bastholt L, Dreno B, Fargnoli MC, Forsea AM, Frenard C, Harwood CAlpha, Hauschild A, Hoeller C, Kandolf-Sekulovic L, Kaufmann R, Kelleners-Smeets NW, Malvehy J, Del Marmol V, Middleton MR, Moreno-Ramirez D, Pellecani G, Peris K, Saiag P, van den Beuken-van Everdingen MHJ, Vieira R, Zalaudek I, Eggermont AMM, Grob JJ; European Dermatology Forum (EDF), the European Association of Dermato-Oncology (EADO) and the European Organization for Research and Treatment of Cancer (EORTC). European interdisciplinary guideline on invasive squamous cell carcinoma of the skin: Part 1. epidemiology, diagnostics and prevention. Eur J Cancer. 2020 Mar;128:60-82. doi: 10.1016/j.ejca.2020.01.007. Epub 2020 Feb 26. PMID 32113941
- [Result] Stratigos AJ, Garbe C, Dessinioti C, Lebbe C, Bataille V, Bastholt L, Dreno B, Concetta Fargnoli M, Forsea AM, Frenard C, Harwood CA, Hauschild A, Hoeller C, Kandolf-Sekulovic L, Kaufmann R, Kelleners-Smeets NWJ, Malvehy J, Del Marmol V, Middleton MR, Moreno-Ramirez D, Pellecani G, Peris K, Saiag P, van den Beuken-van Everdingen MHJ, Vieira R, Zalaudek I, Eggermont AMM, Grob JJ; European Dermatology Forum (EDF), the European Association of Dermato-Oncology (EADO) and the European Organization for Research and Treatment of Cancer (EORTC). European interdisciplinary guideline on invasive squamous cell carcinoma of the skin: Part 2. Treatment. Eur J Cancer. 2020 Mar;128:83-102. doi: 10.1016/j.ejca.2020.01.008. Epub 2020 Feb 26. PMID 32113942
- [Result] Migden MR, Rischin D, Schmults CD, Guminski A, Hauschild A, Lewis KD, Chung CH, Hernandez-Aya L, Lim AM, Chang ALS, Rabinowits G, Thai AA, Dunn LA, Hughes BGM, Khushalani NI, Modi B, Schadendorf D, Gao B, Seebach F, Li S, Li J, Mathias M, Booth J, Mohan K, Stankevich E, Babiker HM, Brana I, Gil-Martin M, Homsi J, Johnson ML, Moreno V, Niu J, Owonikoko TK, Papadopoulos KP, Yancopoulos GD, Lowy I, Fury MG. PD-1 Blockade with Cemiplimab in Advanced Cutaneous Squamous-Cell Carcinoma. N Engl J Med. 2018 Jul 26;379(4):341-351. doi: 10.1056/NEJMoa1805131. Epub 2018 Jun 4. PMID 29863979
- [Result] Porceddu SV, Bressel M, Poulsen MG, Stoneley A, Veness MJ, Kenny LM, Wratten C, Corry J, Cooper S, Fogarty GB, Collins M, Collins MK, Macann AMJ, Milross CG, Penniment MG, Liu HY, King MT, Panizza BJ, Rischin D. Postoperative Concurrent Chemoradiotherapy Versus Postoperative Radiotherapy in High-Risk Cutaneous Squamous Cell Carcinoma of the Head and Neck: The Randomized Phase III TROG 05.01 Trial. J Clin Oncol. 2018 May 1;36(13):1275-1283. doi: 10.1200/JCO.2017.77.0941. Epub 2018 Mar 14. PMID 29537906
- [Result] Harris BN, Pipkorn P, Nguyen KNB, Jackson RS, Rao S, Moore MG, Farwell DG, Bewley AF. Association of Adjuvant Radiation Therapy With Survival in Patients With Advanced Cutaneous Squamous Cell Carcinoma of the Head and Neck. JAMA Otolaryngol Head Neck Surg. 2019 Feb 1;145(2):153-158. doi: 10.1001/jamaoto.2018.3650. PMID 30570645
- [Result] Porceddu SV, Daniels C, Yom SS, Liu H, Waldron J, Gregoire V, Moore A, Veness M, Yao M, Johansen J, Mehanna H, Rischin D, Le QT. Head and Neck Cancer International Group (HNCIG) Consensus Guidelines for the Delivery of Postoperative Radiation Therapy in Complex Cutaneous Squamous Cell Carcinoma of the Head and Neck (cSCCHN). Int J Radiat Oncol Biol Phys. 2020 Jul 15;107(4):641-651. doi: 10.1016/j.ijrobp.2020.03.024. Epub 2020 Apr 11. PMID 32289475
- [Result] Carvalho HA, Villar RC. Radiotherapy and immune response: the systemic effects of a local treatment. Clinics (Sao Paulo). 2018 Dec 10;73(suppl 1):e557s. doi: 10.6061/clinics/2018/e557s. PMID 30540123
- [Result] Bottomley MJ, Thomson J, Harwood C, Leigh I. The Role of the Immune System in Cutaneous Squamous Cell Carcinoma. Int J Mol Sci. 2019 Apr 24;20(8):2009. doi: 10.3390/ijms20082009. PMID 31022866
- [Result] Wild AT, Ye X, Ellsworth SG, Smith JA, Narang AK, Garg T, Campian J, Laheru DA, Zheng L, Wolfgang CL, Tran PT, Grossman SA, Herman JM. The Association Between Chemoradiation-related Lymphopenia and Clinical Outcomes in Patients With Locally Advanced Pancreatic Adenocarcinoma. Am J Clin Oncol. 2015 Jun;38(3):259-65. doi: 10.1097/COC.0b013e3182940ff9. PMID 23648440
- [Result] Kuo P, Bratman SV, Shultz DB, von Eyben R, Chan C, Wang Z, Say C, Gupta A, Loo BW Jr, Giaccia AJ, Koong AC, Diehn M, Le QT. Galectin-1 mediates radiation-related lymphopenia and attenuates NSCLC radiation response. Clin Cancer Res. 2014 Nov 1;20(21):5558-69. doi: 10.1158/1078-0432.CCR-14-1138. Epub 2014 Sep 4. PMID 25189484
- [Result] Pike LRG, Bang A, Mahal BA, Taylor A, Krishnan M, Spektor A, Cagney DN, Aizer AA, Alexander BM, Rahma O, Balboni T, Ott PA, Hodi FS, Schoenfeld JD. The Impact of Radiation Therapy on Lymphocyte Count and Survival in Metastatic Cancer Patients Receiving PD-1 Immune Checkpoint Inhibitors. Int J Radiat Oncol Biol Phys. 2019 Jan 1;103(1):142-151. doi: 10.1016/j.ijrobp.2018.09.010. Epub 2018 Sep 15. PMID 30227198
- [Result] Jarosz-Biej M, Smolarczyk R, Cichon T, Kulach N. Tumor Microenvironment as A "Game Changer" in Cancer Radiotherapy. Int J Mol Sci. 2019 Jun 29;20(13):3212. doi: 10.3390/ijms20133212. PMID 31261963
- [Result] Wysong A, Newman JG, Covington KR, Kurley SJ, Ibrahim SF, Farberg AS, Bar A, Cleaver NJ, Somani AK, Panther D, Brodland DG, Zitelli J, Toyohara J, Maher IA, Xia Y, Bibee K, Griego R, Rigel DS, Meldi Plasseraud K, Estrada S, Sholl LM, Johnson C, Cook RW, Schmults CD, Arron ST. Validation of a 40-gene expression profile test to predict metastatic risk in localized high-risk cutaneous squamous cell carcinoma. J Am Acad Dermatol. 2021 Feb;84(2):361-369. doi: 10.1016/j.jaad.2020.04.088. Epub 2020 Apr 25. PMID 32344066
- [Result] Litchman GH, Fitzgerald AL, Kurley SJ, Cook RW, Rigel DS. Impact of a prognostic 40-gene expression profiling test on clinical management decisions for high-risk cutaneous squamous cell carcinoma. Curr Med Res Opin. 2020 Aug;36(8):1295-1300. doi: 10.1080/03007995.2020.1763283. Epub 2020 May 18. PMID 32372702
- [Result] Farberg AS, Hall MA, Douglas L, Covington KR, Kurley SJ, Cook RW, Dinehart SM. Integrating gene expression profiling into NCCN high-risk cutaneous squamous cell carcinoma management recommendations: impact on patient management. Curr Med Res Opin. 2020 Aug;36(8):1301-1307. doi: 10.1080/03007995.2020.1763284. Epub 2020 May 18. PMID 32351136

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT05246228/Prot_SAP_000.pdf